CLINICAL TRIAL: NCT07072195
Title: A Multicenter, Randomized, Double-Blind, Placebo-controlled, Phase 2 Clinical Trial to Evaluate the Efficacy and Safety of AMC6156 in Patients With Sarcopenia
Brief Title: A Study of AMC6156 in People With Sarcopenia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Animuscure Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMC6156_SP_P2A01
Record Dates: First submitted 2025-07-09; First posted 2025-07-18 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Sarcopenia in Elderly; Sarcopenia
Keywords: sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- AMC6156 0.1mg Treatment Group (Experimental)
  Interventions: Drug: AMC6156 0.1mg
- AMC6156 0.3mg Treatment Group (Experimental)
  Interventions: Drug: AMC6156 0.3mg
- AMC6156 1.0mg Treatment Group (Experimental)
  Interventions: Drug: AMC6156 1.0mg
- Placebo Control Group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AMC6156 0.1mg — Oral administration of AMC6156 in tablet form at a dose of 0.1 mg once daily for 12 weeks.
  Arms: AMC6156 0.1mg Treatment Group
Drug: AMC6156 0.3mg — Oral administration of AMC6156 in tablet form at a dose of 0.3 mg once daily for 12 weeks.
  Arms: AMC6156 0.3mg Treatment Group
Drug: AMC6156 1.0mg — Oral administration of AMC6156 in tablet form at a dose of 1.0 mg once daily for 12 weeks.
  Arms: AMC6156 1.0mg Treatment Group
Drug: Placebo — Oral administration of placebo tablets matching AMC6156 in appearance, once daily for 12 weeks.
  Arms: Placebo Control Group

SUMMARY:
This clinical trial aims to find out whether AMC6156 can improve physical function and is safe in older adults with sarcopenia. Participants will take AMC6156 or a placebo daily for 12 weeks, and their movement, strength, and safety will be regularly monitored through tests and checkups.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation with written informed consent
* Male ≥ 65 years or postmenopausal female
* Diagnosed with sarcopenia:
* ASM < 7.0 kg/m² (men) or < 5.4 kg/m² (women)
* Plus low handgrip strength or SPPB ≤ 9
* MNA screening score ≥ 8
* Body weight ≥ 35 kg, BMI between 15-30 kg/m²
* Willing and able to follow exercise and nutrition guidance

Exclusion Criteria:

* Allergy to investigational drug
* History of GI bleeding, ulcers, or severe liver/kidney/heart disease
* QTc ≥ 450 ms with symptoms
* Severe COPD, uncontrolled diabetes or thyroid disease
* Diseases causing cachexia or muscle wasting (e.g., ALS, Parkinson's)
* Vitamin D deficiency (<10 ng/mL), hemoglobin <10 g/dL
* Severe psychiatric disorders or MMSE < 21
* Inability to walk or recent fracture/surgery affecting mobility
* Use of prohibited medications or recent participation in other clinical trials
* Investigator deems the subject unsuitable for the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in Short Physical Performance Battery (SPPB) Score from Baseline to Week 12 | At Visit 1 (Screening), Visit 2 (Week 0, Baseline), Visit 3 (Week 4), Visit 4 (Week 8), and Visit 5 (Week 12)

SECONDARY OUTCOMES:
Change in Short Physical Performance Battery (SPPB) Score at Week 4 and Week 8 | At Visit 1 (Screening), Visit 2 (Week 0, Baseline), Visit 3 (Week 4), Visit 4 (Week 8), and Visit 5 (Week 12)
Change in Timed Up and Go (TUG) Test Time | At Visit 2 (Week 0), Visit 3 (Week 4), Visit 4 (Week 8), and Visit 5 (Week 12)
Change in Appendicular Skeletal Muscle Mass (ASM) Measured by DXA | At Visit 1 (Screening) and Visit 5 (Week 12)
Change in Handgrip Strength | At Visit 1 (Screening), Visit 2 (Week 0) ,Visit 3 (Week 4), Visit 4 (Week 8), and Visit 5 (Week 12)
Change in SARC-F Score | At Visit 2 (Week 0) and Visit 5 (Week 12)
Change in Sarcopenia Quality of Life (SarQoL) Score | At Visit 2 (Week 0) and Visit 5 (Week 12)

CONTACTS AND LOCATIONS:
Locations (4):
- South Korea (4):
  - CHA Bundang Medical Center, Seongnam-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Seoul National University Hospital, Seoul, Seoul